CLINICAL TRIAL: NCT02439931
Title: Feasibility Study of a Remote Psychosocial Intervention for Brain Tumour Survivors
Brief Title: Remote Psychosocial Intervention for Brain Tumour Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H15-00959
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote psychosocial intervention (Experimental): 10 sessions of remotely delivered psychoeducation and support
  Interventions: Behavioral: Remote psychosocial intervention

INTERVENTIONS:
Behavioral: Remote psychosocial intervention

SUMMARY:
Survivors of high grade brain tumours frequently experience increases in distress, cognitive challenges, and lessened quality of life. At the same time a range of barriers can make it challenging for these individuals to come into the clinic for appropriate psychosocial support. The proposed study is therefore a feasibility study that is designed to develop a manualized, remotely delivered psychosocial intervention for this population and then to test the acceptability, feasibility, apparent efficacy, and areas for improvement of the developed intervention. Further, a remote neuropsychological testing procedure will be developed and implemented and analogous questions will be asked around this procedure.

DETAILED DESCRIPTION:
Purpose

There would be strong value in developing a brief, manualized, remotely delivered, intervention capable of simultaneously improving both emotional well being and cognitive functioning in survivors of malignant brain tumour. The proposed study is designed to test the acceptability, feasibility, apparent efficacy, and areas for improvement of a newly developed intervention designed for this purpose. This investigation is being undertaken as a step toward conducting an randomized clinical trial.

Research Questions

As a feasibility study there will be no hypotheses tested in this study. Instead, the research will be conducted in order to answer the following four questions about the intervention:

1. How acceptable was the intervention?
2. How feasible was the intervention?
3. How much apparent efficacy did the intervention have?
4. How could the involved processes be improved?

Further the following three questions will be asked around the remote neuropsychological testing procedure:

1. How feasible was the remote neuropsychological testing?
2. How valid was the remote neuropsychological testing?
3. How could the neuropsychological testing processes be improved?

Justification

A general justification for the proposed research will be offered below.

Brain tumour survivors demonstrate very high levels of psychopathology. For example, they have been found to exhibit levels of clinical depression that are three times higher than those found in cancer patients overall. This finding is particularly important because symptoms of depression have also been found to be the strongest single predictor of overall quality of life primary in brain tumour survivors.

The cognitive impacts of brain cancer, which are diverse, also have strongly negative effects on quality of life. Impairments in the areas of memory, attention, and executive functioning are the most common cognitive deficits involved.

Despite this depth of suffering, researchers to date have done relatively little work in developing psychologically based interventions that can help to ameliorate these emotional and cognitive sequelae.

More specifically, the remote aspect of this intervention is justified by the fact that this population faces multiple barriers to coming into the clinic for needed psychosocial care, including: geographical isolation; cognitive impairment; driving prohibition; and fatigue. This reality is reflected in the fact that previous researchers have reported facing faced strong challenges in recruiting participants for time consuming intervention studies of this kind in this population. A remote intervention may offer a means of overcoming this barrier to access.

Finally, due to lengthy wait times and other factors, this is also a population that often struggles to receive needed neuropsychological testing in a timely manner. Therefore, there will also be value in validating a brief, remotely delivered neuropsychological testing procedure in this population, above and beyond the role that doing so will play in validating the particular intervention under investigation here.

Objectives

This study has four primary objectives:

1. to develop and deliver a remotely delivered psychosocial intervention to this high needs population
2. to develop a neuropsychological battery that can be remotely delivered to this same population
3. to answer the four questions listed above in regards to the intervention
4. to answer the three questions listed above in regards to the neuropsych assessment process

Research Design

The proposed design will involve a mixed method feasibility study design. A variety of data sources will be used in order to address the 7 research questions listed above. These data sources will include: self report questionnaires; neuropsychological test batteries; fill-in the blank questionnaires; interviews; and focus groups.

6) Statistical Analysis

The included types of quantitative data analysis will be: descriptive statistics; effect sizes; and repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* have a WHO grade 3 or 4 brain tumour
* be under the care of a BC Cancer Agency (BCCA) centre for their brain tumour
* have a Karnofsky Performance Score of 70 or more
* be capable of offering informed consent
* have a high speed internet connection in the home

Exclusion Criteria:

* experiencing levels of distress that will make participation untenable and/or likely counter-productive
* currently experiencing suicidal ideation
* not be capable of speaking English at level such that a translator will be needed to obtain informed consent and/or for the participant to engage appropriately in the intervention/assessments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score on Quality of Life score on the Functional Assessment of Cancer Therapy-Brain | Comparison of scores pre-intervention to immediately post intervention (10 weeks) and 4 month followup
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is a self report measure designed to assess quality of life in people living with brain malignancy across five dimensions: physical well-being, social/family well-being, emotional well being, functional well-being, and disease specific challenges.

SECONDARY OUTCOMES:
Changes in scores regarding psychological distress(anxiety, depression and somatization) on the Brief Symptom Inventory -18 | Comparison of scores pre-intervention to immediately post intervention (10 weeks) and 4 month followup
  The Brief Symptom Inventory -18 is a commonly used self report measure of psychological distress in oncology patients.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas P Ozier, PhD, Principal Investigator — British Columbia Cancer Agency